CLINICAL TRIAL: NCT03465137
Title: Developing a Mechanistic Neurobiological Model of Exposure Therapy Response Based on Fear Extinction Theory
Brief Title: Using the Neuroscience of Fear Extinction for Anxiety Reduction
Acronym: UNFEAR
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: PI left institution
Sponsor: Stanford University (Other)
Responsible Party: Principal Investigator, Tali Manber Ball, PhD, Postdoctoral Scholar, Stanford University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IRB-44722
Record Dates: First submitted 2018-03-07; First posted 2018-03-14 (Actual); Last update posted 2021-10-08 (Actual); Status verified 2021-09

CONDITIONS: Social Anxiety
Keywords: Exposure therapy; Behavioral therapy; fMRI; Extinction learning; Social anxiety
MeSH Terms: interventions — Therapeutics

STUDY DESIGN:
Intervention Model Description: Immediate therapy versus waitlist arms
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Immediate therapy (Experimental): Participants randomized to the immediate therapy arm will receive a weekly individual psychotherapy intervention called Coordinated Anxiety Learning and Management (CALM). The CALM program is an evidence based, exposure-focused therapy (http://calmtoolsforliving.org). Its computer-assisted format guides the therapist through psychoeducation, an introduction to cognitive restructuring, in-session and at-home exposures, and relapse prevention. Therapy will be delivered in 10 weekly 50-minute sessions within a 12 week period.
  Interventions: Behavioral: Coordinated Anxiety Learning and Management (CALM)
- Waitlist (No Intervention): Participants randomized to the waitlist arm will receive no intervention for 12 weeks. After this 12 week period they will receive a the same weekly individual psychotherapy intervention as the immediate therapy group: Coordinated Anxiety Learning and Management (CALM). The CALM program is an evidence based, exposure-focused therapy (http://calmtoolsforliving.org). Its computer-assisted format guides the therapist through psychoeducation, an introduction to cognitive restructuring, in-session and at-home exposures, and relapse prevention. Therapy will be delivered in 10 weekly 50-minute sessions within a 12 week period.

INTERVENTIONS:
Behavioral: Coordinated Anxiety Learning and Management (CALM) — Exposure-focused cognitive behavioral therapy
  Arms: Immediate therapy

SUMMARY:
Social anxiety disorder affects as many as 12% of Americans, resulting in significant distress and disability. Although exposure therapy is one of the best treatments available, as many as 25% of patients do not respond and we do not know why. Extinction learning is thought to be the mechanism of exposure therapy, and the neuroscience of extinction learning has advanced significantly since exposure therapy was developed; however, there has been little application towards improved clinical outcomes.

This project aims to improve exposure therapy response for patients with social anxiety disorder by directly linking exposure therapy response to the neurobiology of extinction learning. It also aims to increase our scientific understanding of how brain circuits work to support extinction learning. To do this, 80 adults with social anxiety disorder will randomly be assigned to either receive exposure therapy right away, or to wait before therapy. Participants will all complete a functional magnetic resonance imaging scan to assess extinction learning before the therapy.

DETAILED DESCRIPTION:
The best available treatment for social anxiety disorder is exposure therapy; however, 25% of socially anxious patients do not respond to an adequate course of exposure therapy and it is unclear why. Prior attempts to identify non-responders using clinical and demographic features have been largely unsuccessful, highlighting the need to examine constructs that are more closely tied to the mechanism of treatment (i.e., extinction learning and recall) and the organ of dysfunction (i.e., the brain). The neurobiology of extinction learning and recall is well understood from decades of animal and pre-clinical laboratory work, which has highlighted the importance of the amygdala, dorsal anterior cingulate cortex (dACC), and ventromedial prefrontal cortex (vmPFC). However, this knowledge has not been leveraged to improve exposure therapy response, despite the assumption that response relies on extinction learning and its successful recall.

Thus, a critical long-term goal is to improve exposure therapy response by tailoring therapy based on the neurobiological profile of each patient. This project addresses that goal by directly linking neurobiological profiles of extinction learning and recall with clinical symptoms and therapy response. A major objective of this project is therefore to build a mechanistic predictive model of exposure therapy response based on the neurobiology of extinction learning and recall.

To accomplish this goal, the investigators will recruit 80 adults with social anxiety disorder who will be randomized to 10 sessions of exposure-focused therapy or waitlist. The primary clinical outcome measure will be the Liebowitz Social Anxiety Scale (LSAS), a validated and widely used measure that assesses anxiety and avoidance symptoms. Pre-therapy, participants will also undergo an experimental protocol for extinction learning and recall. Participants will first view a neutral abstract image repeatedly paired with a loud aversive noise, and another image that is never paired (fear acquisition phase). Following this, participants will view the same images without aversive consequences (extinction learning phase). Better extinction learning will be defined as greater reductions in skin conductance within the extinction learning phase. Brain activation during extinction learning will be assessed in the amygdala, dACC, and vmPFC. Finally, participants will view the same images without aversive consequences one week later (extinction recall phase). Better extinction recall will be defined as less skin conductance during extinction recall relative to fear acquisition. The central hypothesis is that greater activation in the vmPFC during extinction learning will predict both extinction recall and therapy response over and above symptom severity.

ELIGIBILITY:
Inclusion Criteria:

* age 18-50
* primary diagnosis of social anxiety disorder
* fluent spoken and written English
* able to provide informed consent.

Exclusion Criteria:

* history of mania or psychosis
* current moderate or severe substance use disorder
* current major depression greater than moderate severity
* high risk for suicide
* prior traumatic brain injury with loss of consciousness >5 minutes
* general medical condition or impediment to vision, hearing, or motor function likely to interfere with assessments
* prior exposure therapy (>2 sessions)
* current use of psychotropic medication
* current psychotherapy other than couples counseling
* post-menopausal status
* pregnancy

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 32 (Actual)
Dates: Start 2018-01-14 (Actual); Primary Completion 2021-09-30 (Actual); Study Completion 2021-09-30 (Actual)

PRIMARY OUTCOMES:
Liebowitz Social Anxiety Scale (LSAS) | 12 weeks
  A validated, widely-used measure of social anxiety severity, with anxiety and avoidance subscales. Subscales range from 0 to 72, with higher scores indicating greater anxiety and avoidance symptoms. A total score is computed by summing the two subscales (range: 0 to 144, higher scores indicate greater social anxiety severity).

SECONDARY OUTCOMES:
Patient Health Questionnaire (PHQ-9) | 12 weeks
  A validated and widely-used measure of depression symptom severity, ranging from 0 to 27, with higher scores indicating greater depression severity.
Brief Fear of Negative Evaluation (BFNE) | 12 weeks
  A validated measure of fear of negative evaluation, a key concept in social anxiety disorder, ranging from 0 to 32, with higher scores indicating greater fear of negative evaluation.
World Health Organization Quality of Life scale (WHO-QOL) | 12 weeks
  A validated measure of quality of life, which has subscales for physical health, psychological health, social relationships, and environment. Subscales scores are each transformed into a 0-100 range, with higher scores indicating better quality of life. There is no total score and the subscales are not combined.

CONTACTS AND LOCATIONS:
Locations (1):
- Stanford University Department of Psychiatry & Behavioral Sciences, Palo Alto, California, United States

IPD SHARING:
Plan to Share IPD: Yes
We plan to voluntarily share the raw fMRI data generated by this project through openfmri.org, a project of the Stanford Center for Reproducible Neuroscience. OpenfMRI is a recommended repository for several academic journals. There is no cost for researchers or analysts for use of this repository; the OpenfMRI repository uses a Public Domain license. We will fully de-identify and anonymize our data before uploading to the database, consistent with the OpenfMRI policy. Furthermore, the purpose, risks, and benefits of data sharing will be included in our consent form, and participants will be given the opportunity to exclude their data from the repository. Only participants who consent to and provide HIPAA authorization for this use will have their data uploaded.
Time Frame: We anticipate uploading the final research data of all consenting participants no later than 5 years after the completion of the study.